CLINICAL TRIAL: NCT00426595
Title: Pharmacokinetics of Enteral Omeprazole Suspension in Patients With Cerebral Palsy and Mental Retardation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Myriam Van Winckel, University Hospital Ghent
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2007/013
Record Dates: First submitted 2007-01-23; First posted 2007-01-25 (Estimated); Last update posted 2009-04-10 (Estimated); Status verified 2009-04

CONDITIONS: Gastreoesophageal Reflux Disease

INTERVENTIONS:
Drug: Administration of omeprazole suspension
Drug: omeprazole administered as a multi-unit-pellet system

SUMMARY:
Gastroesophageal reflux disease and reflux-esophagitis are a major chronic problem in most children with cerebral palsy and mental retardation. Oral administration of enteric-coated formulations of the acid-labile proton pump inhibitor omeprazole is often problematic in these patients who may be suffering from swallowing disorders. A suspension of omeprazole in a sodium bicarbonate solution is often used for administration via the gastrostomy tube. This trial aims to compare the pharmacokinetics of omeprazole administered through the gastrostomy tube as a suspension in pediatric patients with cerebral palsy and mental retardation versus the pharmacokinetics of omeprazole administered as a multi-unit-pellet system (MUPS®). The crossover study will consist of 2 consecutive treatment periods of 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Children > 15 kg
* Cerebral palsy and mental retardation with swallowing disorders
* Presence of gastrostomy tube
* GERD and/or reflux-esophagitis treated with omeprazole at the same dose since at least 2 weeks
* Informed consent

Exclusion Criteria:

* Treatment with ciclosporine, tacrolimus, mycofenolate
* Treatment with anticoagulants
* Infection
* Recent start of treatment with known inhibitors of the omeprazole-metabolism
* Moderate to severe hepatic impairment (SGPT and/or AST > 3 times upper limit)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Estimated)
Dates: Start 2007-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (at the end of the treatment period of 14 days)

SECONDARY OUTCOMES:
Gastric pH (at the end of the treatment period of 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Myriam Van Winckel, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be